CLINICAL TRIAL: NCT05311332
Title: Assessment of Horizontal Bone Gain Using Computer-guided vs. Conventional Cortical Shell Technique for Horizontal Maxillary Alveolar Ridge Augmentation
Brief Title: Computer-guided vs. Conventional Cortical Shell Technique for Horizontal Augmentation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Future University in Egypt (Other)
Responsible Party: Principal Investigator, Dina Ayman, assistant lecturer, Future University in Egypt
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FUE.REC (23)\11-2021
Record Dates: First submitted 2022-03-27; First posted 2022-04-05 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Alveolar Bone Resorption; Horizontal Ridge Deficiency
Keywords: alveolar ridge deficiency; computer guided surgery; chin graft

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anterior maxillary bone augmentation using computer guided autogenous cortical shell technique. (Experimental): a patient-specific guide was used to harvest a chin cortical shell which was also prepared and positioned at the (anterior horizontally atrophied maxilla) recipient site using another patient-specific positioning guide.
  Interventions: Procedure: Augmentation of horizontal deficient anterior maxilla with a cortical shell harvested from a chin using patient specific surgical guide then positioned with another guide
- Anterior maxilla bone augmentation using free hand autogenous cortical shell technique. (Active Comparator): the horizontally atrophic anterior maxilla was augmented with a cortical shell technique the bone was harvested from the chin without a patient-specific guide.
  Interventions: Procedure: Augmentation of horizontal deficient anterior maxilla with a cortical shell harvested from a chin

INTERVENTIONS:
Procedure: Augmentation of horizontal deficient anterior maxilla with a cortical shell harvested from a chin — Augmentation of horizontal deficient anterior maxilla using the conventional protocol of cortical shell technique
  Arms: Anterior maxilla bone augmentation using free hand autogenous cortical shell technique.
Procedure: Augmentation of horizontal deficient anterior maxilla with a cortical shell harvested from a chin using patient specific surgical guide then positioned with another guide — using a patient-specific surgical guide to harvest bone cortical shell from the chin and another patient-specific surgical guide to fix it in the atrophied maxillary anterior area
  Arms: Anterior maxillary bone augmentation using computer guided autogenous cortical shell technique.

SUMMARY:
this study aims to evaluate horizontal bone augmentation achieved at the anterior maxilla using computer-guided cortical shell bone technique and accuracy of fixation of the bone shell away from the atrophic ridge by a calculated distance which is always a challenging step for inexperienced surgeons to fix a cortical shell at the ideal position in the conventional protocol it was never guided to be precisely fixed at the proper position and angulation the problem is if it fixed with insufficient distance with proposed volume loss leads to totally insufficient volume gain for future implant placement also to evaluate the efficacy of the CAD/CAM surgical guide during chin harvesting procedures in reducing the risk of anatomical structure damage and patient morbidity with more accuracy compared with the standard technique. this trial versus free hand conventional cortical shell bone technique both harvested from symphysis area (chin).

DETAILED DESCRIPTION:
Tooth extraction may be due to a variety of causes such as badly decayed, periodontal disease, and trauma whatever the reason tooth loss is always followed by loss of masticatory force and muscle stimulation to the alveolar bone so according to Wolff's Law (Wolff, 1892) loss of mechanical stimulation is followed by the reduction of bone mass.

Several surgical protocols have been used to manage horizontal maxillary alveolar bone atrophy such as bone splitting and bone spreading techniques with or without filling the created space, onlay bone graft, guided bone regeneration using resorbable or non-resorbable membrane, distraction osteogenesis, and shell bone block technique which use a thin cortical bone shell to reshape the atrophied ridge and protect the particulate bone graft.

Despite the popularity of this technique, it usually requires high surgical skills, prolonged intra-operative time, and unfortunately has some technical drawbacks. Such as lack of anatomical guidance during bone harvesting which may lead to injury to the important vital structure and lack of guidance during fixation may lead to improperly positioned, tilted, or rotated shell or even leaving an undesired distance between the shell and deficient ridge

With the increasing use of cone-beam computed tomography (CBCT), intra and extra oral scanner for patient data acquisition, and complete digital workflow in clinical practice and it is rapidly becoming the standard of care in dentistry. Regarding bone augmentation as preparation for future implant placement. computer-aided surgery has been an innovation that enables clinicians to have firm and accurate treatment planning. Also, milling or 3D printing methods allow variable techniques for the fabrication of surgical templates.

This study aims to fully digitalize such technique using patient-specific surgical guides to allow for accurate graft harvesting and positioning and to minimize intraoperative time and complications associated with this procedure

ELIGIBILITY:
Inclusion Criteria:

* patient free from any systemic condition.
* Edentulous anterior maxilla with a horizontal deficient alveolar ridge that is less than 4 mm measured from outer buccal cortices to outer palatal cortices.
* Highly motivated patients are willing for the surgical procedure and follow-up, with informed consent.

Exclusion Criteria:

* Intra bony lesions (e.g. Cysts) or infections(e.g.abcess) that may retard the osteotomy healing.
* Medically compromised patients.
* Uncooperative patients.
* Patients with any diseases or taking any medications that compromise bone healing

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2021-10-13 (Actual); Primary Completion 2022-08-20 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
Alveolar ridge horizontal net bone gain | 4 months
  volumetric change of deficient alveolar ridge after augmentation

SECONDARY OUTCOMES:
surgical procedure accuracy | immediate post operative
  depening on the superimposition between immediate postoperative CBCT scan over planning
intraoperation time | at time of surgery
  duration of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Dina Ayman Fayek, BDS, Principal Investigator — teaching assistant oral and maxillofacial department future university in Egypt
Locations (1):
- future university in Egypt, faculty of dentistry, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
the data will be available from the corresponding author upon resonable request.

REFERENCES:
- [Derived] Ayman D, Shawky M, Aly LAA, Mounir M, Zekry AKA. Bone gain and accuracy assessment of computer-guided workflow for horizontal augmentation of atrophic anterior maxilla with symphyseal cortical plates: a randomized controlled trial. BMC Oral Health. 2025 Jul 2;25(1):1039. doi: 10.1186/s12903-025-06415-2. PMID 40604890